CLINICAL TRIAL: NCT02491931
Title: Oral Glutamine Reduces Myocardial Damage After Coronary Revascularization Under Cardiopulmonary Bypass
Brief Title: Oral Glutamine in Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, MD., Ph.D., F.A.C.S., Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Glutamine-2015
Record Dates: First submitted 2015-06-23; First posted 2015-07-08 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Heart Disease
Keywords: Cardiac Surgical Procedures; Cardiovascular Surgical Procedures; Dietary Supplements; Glutamine; TROPONIN I; cardiopulmonary bypass
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLN group (Active Comparator): All patients in the GLN group received an oral GLN supplement. The total GLN dose given to patients was standardized to 0.5 g/kg/day during 3 days prior to CPB, and one final dose of 0.25 g/kg/day of GLN/maltodextrin in the morning of surgery 4 hours prior to initiation of anesthesia.
  Interventions: Dietary Supplement: Supplement/placebo intake
- CONT group (Placebo Comparator): All patients in the GLN group received an oral maltodextrin supplement, similar in shape and texture as GLN supplement. The total placebo given to patients was standardized to 0.5 g/kg/day during 3 days prior to CPB, and one final dose of 0.25 g/kg/day of maltodextrin in the morning of surgery 4 hours prior to initiation of anesthesia.
  Interventions: Dietary Supplement: Supplement/placebo intake

INTERVENTIONS:
Dietary Supplement: Supplement/placebo intake — Patients will receive either GLN or placebo prior to cardiovascular surgery under extracorporeal circulation, during 3 days and one final dose 4 hours prior to anesthesia.

SUMMARY:
Introduction: Glutamine (GLN) is the most abundant free amino acid in the body. It modulates immune cell function and is an important energy substrate for most cells (especially for enterocytes and lymphocytes) in critical patients. GLN levels significantly decreased during sepsis/critical illness leading to an increase in infectious complications, organ failure and mortality. Moreover, in cases of ischemia/reperfusion injury in the myocardium, GLN increases the levels of Adenosine triphosphate (ATP)/Adenosine diphosphate (ADP) ratio and prevents intracellular lactate accumulation. Recently, the perioperative effect of intravenous and oral GLN treatment been associated in lowering levels of cardiac injury markers such as Troponin-I (TROP-I) and the number of postoperative complications in patients who underwent Cardiopulmonary Bypass (CPB). The aim of the study was to analyze the oral dose of preoperative oral GLN treatment in patients who underwent CPB with extracorporeal circulation in Mexican patients.

DETAILED DESCRIPTION:
INTRODUCTION Glutamine (GLN) is the most abundant free amino acid in the body, and commonly known as a non-essential amino acid due to the ability of most cells to produce it. It has many essential metabolic functions in the organism; it is an energy substrate for most cells (especially for enterocytes and lymphocytes), a precursor for nucleotide, glutamate, and (in particular) glutathione synthesis, and an important cellular antioxidant. It plays a central role in nitrogen transport within the body, and is the most important substrate for renal ammoniagenesis.

Studies have demonstrated that the presence of GLN in the medium regulates glutamine synthetase expression via a post-transcriptional mechanism, where the rate of glutamine synthetase protein degradation is diminished and its activity, augmented, in the presence of low GLN concentration. This amino acid modulates immune cell function and production of cytokines via attenuation of multiple pathways of inflammation, such as Nuclear Factor kB (NF-kB), protein kinases, inhibition of increases in Nitric Oxide Synthase (iNOS) expression.

It has been shown to be beneficial for the metabolically stressed patient, especially the critically ill patients. During acute illnesses, patients experience nutritional depletion, which correlates with low plasma and low mucosal GLN concentrations.

GLN levels are significantly decreased in critical illness, leading to an increase in infectious complications, organ failure and mortality. Moreover, in cases of ischemia/reperfusion injury, GLN increases the myocardial ATP/ADP ratio and prevents intracellular lactate accumulation.

GLN has been shown to be a key nutrient in the body's response to stress and injury described in multiple studies with in vitro and in vivo myocardial injury following I/R. These include enhanced myocardial glutathione, adenosine triphosphate (ATP), and glutamate (a major stress substrate for the stressed myocardium) post-I/R injury, and induction of heat shock proteins, especially Heat Shock Protein-70 (HSP-70) in critically ill patients. The stress tolerance provided by HSP-70 can protect against cellular injury, lung injury, ischemia/reperfusion injury, and septic shock, by the GLN influences on the inflammatory response, oxidative stress, apoptosis modulation, and the integrity of gut barrier.

Protection of the myocardium following ischemia and reperfusion injury is crucial in the perioperative management of patients after cardiopulmonary bypass (CPB). This ischemia is the most important factor of reversible perioperative risk for cardiovascular complications. Patients undergoing CPB with a heart-lung machine (termed cardiopulmonary bypass) are at an increased risk of having abnormal "inflammation" in their body after surgery. Such inflammation can contribute to slower recovery from surgery, an increased risk of infection, an increased risk of damage to organs other than the heart, and a more complicated course.

Numerous experimental and clinical trials have demonstrated the cardioprotective effects of GLN, including dose-dependent enhanced myocardial functional recovery following acute normothermic ischemia in the rat. GLN has also been shown to reduce infarct size to approximately 39% in a rabbit model following ischemia/reperfusion injury.[19] GLN treatment also increased load tolerance in patients with ischemic heart disease (IHD).

In 2012, a clinical study observed a significant decrease in TROP-I in patients with ischemic heart disease who underwent CPB with extracorporeal circulation who received (0.4 g/kg of GLN, Dipeptiven solution) one day before surgery. The case group (n=25) showed reduced levels of TROP-I compared to control group (1.2 ng/ml to 2.4 ng/ml), p=0.035 on the first postoperative day. Also, the median cardiac index and median stroke index were higher in case group following CPB, improving myocardial function.

In another study, the authors observed significantly decreased TROP-I levels in their pilot-clinical trial. They performed an oral intervention in patients undergoing CPB, giving 25 g twice of GLN supplement. TROP-I levels were significantly lower at 24, 48, and 72 postoperatively hours (all p < 0.05).

Despite the varied experimental data showing the cardioprotective effects of GLN, there is a lack of clinical trials with CPB patients. The finding that lower levels of cardiac injury markers are observed in patients treated with oral GLN prior to CPB can have major implications in these patients. The purpose of this study is to analyze the effect of a preoperative oral supplementation of GLN in reducing postoperative levels of Troponin-I in Mexican patients who underwent CPB under extracorporeal circulation. The oral GLN proposed in this study is based on what has been previously studied and what is considered safe.

MATERIALS AND METHODS. A controlled clinical trial performed in 28 patients who underwent cardiopulmonary bypass with confirmed diagnosis of ischemic heart disease. The protocol was made between January 2013 and December 2014 in the Specialty Hospital of the Western National Medical Center, Mexican Institute of Social Security.

The protocol received ethics approval by the Local Committee of Ethics in Research and Health. All patients gave informed consent prior to participation.

Participants were men or nonpregnant women, aged 40-70 years. Participants were excluded on the basis of preexisting kidney, liver dysfunction or other comorbid conditions such as drug or alcohol abuse, positivity to human immunodeficiency virus (HIV), hepatitis B / C or allergies against components of GLN. Participants were also excluded on the basis of signs of ongoing ischemia, defined by persistent elevation of TROP-I and CK-MB levels. They were also excluded if they were on a diet with any supplemental GLN.

Treatment Following study enrollment, patients were randomized (blinded envelopes that were opened sequentially by a blinded study pharmacist), to receive either oral GLN supplement group or control group (CONT) with maltodextrin (as isocaloric complex carbohydrate).

All investigators and clinical caregivers were blinded to study intervention. All patients in the GLN group received a GLN supplement. The total GLN/maltodextrin dose given to patients was standardized to 0.5 g/kg/day during 3 days prior to CPB, and taking one final dose of 0.25 g/kg/day of GLN/maltodextrin in the morning of surgery 4 hours prior to initiation of anesthesia.

Compliance with ingestion of the study drug was assessed via daily reminder calls from the study investigator and required empty package returns.

Patient Sample Collection and Analysis Blood was collected at baseline (one hour before surgery), and then one hour after surgery and 12 and 24 postoperative hours. After collection, blood was processed for analysis of cardiac injury markers: TROP-I, creatine phosphokinase (CPK) and creatine phosphokinase-Mb (CPK-Mb) and were analyzed using Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD).

Clinical Data Collection All patients had essential demographic information collected as well as preoperative cardiac ejection fraction at study enrollment. In addition, postoperative complications were evaluated, including stroke, infections and postoperative vasopressor therapy. The time of time of aortic clamp during surgery and days in the Critial Care Unit (UCI) were measured. Mortality in the postoperative period was also collected.

Statistical Analysis Qualitative variables are expressed as raw numbers and proportions, whereas the quantitative variables are expressed as means ± standard deviations. To compare quantitative variables in the the results between the two groups, the U Mann Whitney test was used. Qualitative variables were measured using Chi 2 of Fisher's exact test in any expected values below 5. A p value of 0.05 or less was considered significant. The analysis was performed using Excel 2013 and Statistical Package for the Social Sciences (SPSS) version 20 for Windows (IBM Corp., NY, USA).

Ethical Considerations The study was conducted according to the principles of the Declaration of Helsinki and the Guidelines for Health Research in Mexico. The protocol was approved by the Local Committee on Health Research.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of Ischemic heart disease in whom cardiac revascularization (cardiac by pass) was going to be performed.
* Written informed consent from each patient.

Exclusion Criteria:

* Preexisting kidney disease
* Liver dysfunction

  .Drug or alcohol abuse Positivity to human immunodeficiency virus (HIV)
* Hepatitis B / C
* Allergies against components of GLN.
* Patients with an ongoing ischemia, defined by persistent elevation of TROP-I and CPK-MB levels.
* If any dietetic supplement of GLN was taken simultaneously.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Troponin-I | 1 hour before surgery.
  Blood sample (10 ml) was taken from patient and analyzed to obtain Troponin-I levels were captured using Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD).
Creatine Kinase | 1 hour before surgery
  Blood sample (10 ml) was taken from patient and analyzed to obtain Creatine Kinase levels were captured using Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD).
Creatine Kinase - Mb | 1 hour before surgery
  Blood sample (10 ml) was taken from patient and analyzed to obtain Creatine Kinase-Mb levels were captured using Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD).
Troponin-I | one hour after surgery.
  Blood sample (10 ml) was taken from patient and analyzed to obtain Troponin-I levels were captured using Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD).
Creatine Kinase | one hour after surgery.
  Blood sample (10 ml) was taken from patient and analyzed to obtain Creatine Kinase-Mb levels were captured using Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD).
Creatine Kinase - Mb | one hour after surgery.
  Blood sample (10 ml) was taken from patient and analyzed to obtain Creatine Kinase-Mb levels were captured using Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD).
Troponin-I | 12 hours after surgery
  Blood sample (10 ml) was taken from patient and analyzed to obtain Troponin-I levels were captured using Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD).
Creatine Kinase | 12 hours after surgery
  Blood sample (10 ml) was taken from patient and analyzed to obtain Troponin-I levels were captured using Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD).
Creatine Kinase - Mb | 12 hours after surgery
  Blood sample (10 ml) was taken from patient and analyzed to obtain Troponin-I levels were captured using Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD).
Troponin-I | 24 hours after surgery
  Blood sample (10 ml) was taken from patient and analyzed to obtain Troponin-I levels were captured using Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD).
Creatine Kinase | 24 hours after surgery
  Blood sample (10 ml) was taken from patient and analyzed to obtain Troponin-I levels were captured using Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD).
Creatine Kinase - Mb | 24 hours after surgery
  Blood sample (10 ml) was taken from patient and analyzed to obtain Troponin-I levels were captured using Meso Scale technology (Meso Scale Discovery, Gaithersburg, MD).

SECONDARY OUTCOMES:
Postoperative Stroke | 15 days after surgery.
  Any stroke occurred in patients durin UCI stay was counted as 1 per event, measured in frequency of occurrence.
Length of stay in UCI. | 15 days after surgery.
  The total time of stay in UCI was measured in days in both groups.
Mortality | 15 days after surgery.
  All deceases were captured in both groups during UCI stay until discharge of the patient.
Postoperative Infections | 15 days after surgery.
  Any infections occurred in patients durin UCI stay was counted as 1 per event, measured in frequency of occurrence.
Postoperative vasopressor therapy | 15 days after surgery.
  When any vasopressor was needed during UCI stay, was counted as 1 per event, measured in frequency of occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: González-Ojeda Alejandro, MD. PhD. F.A.C.S., Study Director — Instituto Mexicano del Seguro Social; Chávez-Tostado Mariana, M.Sc. R. Nutr., Principal Investigator — Instituto Mexicano del Seguro Social

REFERENCES:
- [Result] Oliveira GP, Dias CM, Pelosi P, Rocco PR. Understanding the mechanisms of glutamine action in critically ill patients. An Acad Bras Cienc. 2010 Jun;82(2):417-30. doi: 10.1590/s0001-37652010000200018. PMID 20563423
- [Result] Wernerman J. Glutamine supplementation. Ann Intensive Care. 2011 Jul 18;1(1):25. doi: 10.1186/2110-5820-1-25. PMID 21906372
- [Result] Singleton KD, Beckey VE, Wischmeyer PE. GLUTAMINE PREVENTS ACTIVATION OF NF-kappaB AND STRESS KINASE PATHWAYS, ATTENUATES INFLAMMATORY CYTOKINE RELEASE, AND PREVENTS ACUTE RESPIRATORY DISTRESS SYNDROME (ARDS) FOLLOWING SEPSIS. Shock. 2005 Dec;24(6):583-9. doi: 10.1097/01.shk.0000185795.96964.71. PMID 16317391
- [Result] Wischmeyer PE. Glutamine: role in critical illness and ongoing clinical trials. Curr Opin Gastroenterol. 2008 Mar;24(2):190-7. doi: 10.1097/MOG.0b013e3282f4db94. PMID 18301270
- [Result] Coeffier M, Dechelotte P. The role of glutamine in intensive care unit patients: mechanisms of action and clinical outcome. Nutr Rev. 2005 Feb;63(2):65-9. doi: 10.1111/j.1753-4887.2005.tb00123.x. PMID 15762090
- [Result] Oudemans-van Straaten HM, Bosman RJ, Treskes M, van der Spoel HJ, Zandstra DF. Plasma glutamine depletion and patient outcome in acute ICU admissions. Intensive Care Med. 2001 Jan;27(1):84-90. doi: 10.1007/s001340000703. PMID 11280678
- [Result] Jimenez Jimenez FJ, Cervera Montes M, Blesa Malpica AL; Metabolism and Nutrition Working Group of the Spanish Society of Intensive Care Medicine and Coronary units. Guidelines for specialized nutritional and metabolic support in the critically-ill patient: update. Consensus SEMICYUC-SENPE: cardiac patient. Nutr Hosp. 2011 Nov;26 Suppl 2:76-80. doi: 10.1590/S0212-16112011000800017. PMID 22411526
- [Result] Fuentes-Orozco C, Anaya-Prado R, Gonzalez-Ojeda A, Arenas-Marquez H, Cabrera-Pivaral C, Cervantes-Guevara G, Barrera-Zepeda LM. L-alanyl-L-glutamine-supplemented parenteral nutrition improves infectious morbidity in secondary peritonitis. Clin Nutr. 2004 Feb;23(1):13-21. doi: 10.1016/s0261-5614(03)00055-4. PMID 14757388
- [Result] Sufit A, Weitzel LB, Hamiel C, Queensland K, Dauber I, Rooyackers O, Wischmeyer PE. Pharmacologically dosed oral glutamine reduces myocardial injury in patients undergoing cardiac surgery: a randomized pilot feasibility trial. JPEN J Parenter Enteral Nutr. 2012 Sep;36(5):556-61. doi: 10.1177/0148607112448823. Epub 2012 May 23. PMID 22623413
- [Result] Lomivorotov VV, Efremov SM, Shmirev VA, Ponomarev DN, Lomivorotov VN, Karaskov AM. Glutamine is cardioprotective in patients with ischemic heart disease following cardiopulmonary bypass. Heart Surg Forum. 2011 Dec;14(6):E384-8. doi: 10.1532/HSF98.20111074. PMID 22167767
- [Result] Wischmeyer PE, Jayakar D, Williams U, Singleton KD, Riehm J, Bacha EA, Jeevanandam V, Christians U, Serkova N. Single dose of glutamine enhances myocardial tissue metabolism, glutathione content, and improves myocardial function after ischemia-reperfusion injury. JPEN J Parenter Enteral Nutr. 2003 Nov-Dec;27(6):396-403. doi: 10.1177/0148607103027006396. PMID 14621120
- [Result] Groening P, Huang Z, La Gamma EF, Levy RJ. Glutamine restores myocardial cytochrome C oxidase activity and improves cardiac function during experimental sepsis. JPEN J Parenter Enteral Nutr. 2011 Mar;35(2):249-54. doi: 10.1177/0148607110383040. PMID 21378254
- [Result] Villar J, Edelson JD, Post M, Mullen JB, Slutsky AS. Induction of heat stress proteins is associated with decreased mortality in an animal model of acute lung injury. Am Rev Respir Dis. 1993 Jan;147(1):177-81. doi: 10.1164/ajrccm/147.1.177. PMID 8420414
- [Result] Ziegler TR, Ogden LG, Singleton KD, Luo M, Fernandez-Estivariz C, Griffith DP, Galloway JR, Wischmeyer PE. Parenteral glutamine increases serum heat shock protein 70 in critically ill patients. Intensive Care Med. 2005 Aug;31(8):1079-86. doi: 10.1007/s00134-005-2690-5. Epub 2005 Jun 23. PMID 15973519
- [Result] Khogali SE, Harper AA, Lyall JA, Rennie MJ. Effects of L-glutamine on post-ischaemic cardiac function: protection and rescue. J Mol Cell Cardiol. 1998 Apr;30(4):819-27. doi: 10.1006/jmcc.1998.0647. PMID 9602431
- [Result] Twerenbold R, Reichlin T, Reiter M, Muller C. High-sensitive cardiac troponin: friend or foe? Swiss Med Wkly. 2011 May 10;141:w13202. doi: 10.4414/smw.2011.13202. eCollection 2011. PMID 21557113
- [Result] McGuinness J, Neilan TG, Cummins R, Sharkasi A, Bouchier-Hayes D, Redmond JM. Intravenous glutamine enhances COX-2 activity giving cardioprotection. J Surg Res. 2009 Mar;152(1):140-7. doi: 10.1016/j.jss.2008.03.045. Epub 2008 Apr 28. PMID 18708191
- [Result] Khogali SE, Pringle SD, Weryk BV, Rennie MJ. Is glutamine beneficial in ischemic heart disease? Nutrition. 2002 Feb;18(2):123-6. doi: 10.1016/s0899-9007(01)00768-7. PMID 11844641